CLINICAL TRIAL: NCT01086241
Title: A Study to Determine Patient Benefit of Tomosynthesis in Screening Mammography
Brief Title: Tomosynthesis in Screening Mammography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: DX-TOM-001 25232; DX-TOM-001 25232
Record Dates: First submitted 2010-03-11; First posted 2010-03-15 (Estimated); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Breast Density
Keywords: Tomography; Mammography; Breast Neoplasms; Prevention and Control
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: routine 2D mammogram (Active Comparator): Subject receives regular 2D mammogram.
  Interventions: Procedure: 2D Mammogram
- B: Routine Mammogram + tomosynthesis (Active Comparator): Routine Mammogram and tomosynthesis
  Interventions: Procedure: Tomosynthesis

INTERVENTIONS:
Procedure: 2D Mammogram — Those patients randomized to the mammogram arm will receive a regular 2D mammogram. Compression lasts several seconds in order to obtain 4 views. The x-ray tube is programmed to obtain an arc of low dose projection images through the breast.
  Arms: A: routine 2D mammogram
Procedure: Tomosynthesis — Those patients randomized to the tomosynthesis arm will receive a combination of 3D and 2D screening mammogram. The additional tomosynthesis data is obtained immediately after acquisition of the 2D study, with the patient and breast remaining in the same position and compression. Compression lasts about 7 seconds longer for each of the 4 views. The x-ray tube is programmed to obtain an arc of low dose projection images through the breast.
  Arms: B: Routine Mammogram + tomosynthesis

SUMMARY:
Tomosynthesis is a new digital mammographic tool which can be performed at the same time as routine screening mammography. It creates CT-like slices through the breast, minimizing the tissue overlap. Tomosynthesis has the potential to improve screening mammography outcomes by increasing cancer detection rates, decreasing false negative rates and false positive rates. This trial will help determine if tomosynthesis is useful in a screening setting.

DETAILED DESCRIPTION:
We will evaluate the effect of tomosynthesis mammography outcomes in a screening setting. We will collect data on interpretation time, recall rates, cancer detection rates, and interval cancer rates in dense breasts(≥ 50% glandular density). If the interpretation time is less than 4X a routine read, and the recall rates have dropped < 30% of initial values, we will then conduct a study with larger numbers to better evaluate cancer detection rates and interval cancer rates.

ELIGIBILITY:
Inclusion Criteria:

* Females 40-69 years of age attending Screen Test Kingsway referred for a screening mammogram as defined by Canadian Cancer Society guidelines.
* Prior mammogram report indicating ≥ 25% breast density.

Exclusion Criteria:

* Prior mammogram report indicating <25% breast density.
* Breast implants
* Pregnancy

Ages: 40 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2010-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Interpretation Time of Scan | Within 1 month of receiving scan

SECONDARY OUTCOMES:
Recall Rates | 6 month intervals for 2 years after initial scan
Discomfort Scale | Immediately after the subject receives scan

CONTACTS AND LOCATIONS:
Overall Officials: Aalo Bistritz, MD, Study Chair — Cross Cancer Institute; Aalo Bistritz, MD, Principal Investigator — Cross Cancer Institute
Locations (1):
- Alberta Screen Test, Edmonton, Alberta, Canada